CLINICAL TRIAL: NCT06642831
Title: Polycystic Ovarian Syndrome (PCOS) in Human Adolescent and Young Adult Females - Biomarker Evaluation Study (PHOEBE)
Brief Title: Polycystic Ovarian Syndrome (PCOS) Biomarker Evaluation Study
Acronym: PHOEBE
Status: Recruiting | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Collaborators: Roche Diagnostics International AG (Industry)
Responsible Party: Principal Investigator, Laura Lotz, PD Dr. med., University Hospital Erlangen
Other Study IDs: 22-114-B
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
Keywords: PCOS; biomarker; adolescents
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Women with PCOS: Women in the age range of 15-25 years fulfilling the PCOS criteria defined by the International Evidence-based Guideline
- Women without PCOS (controls): Women in the age range of 15-25 years who are negative for the diagnostic criteria of PCOS according to the International Evidence based guideline

SUMMARY:
The purpose of the study is to validate recently identified biomarkers for the identification of PCOS in adolecent and young adult women.

DETAILED DESCRIPTION:
The purpose of the study is to validate potential biomarkers for the aid in the diagnosis of PCOS in adolescent and young adult women in the age range of 15-25 years. Female subjects included in this study will have one visit where clinical data for assessing PCOS will be collected and a blood draw will be performed to collect serum for measurement of parameters relevant to PCOS will be performed. Study subjects that receive a PCOS diagnosis will have two follow up visits for follow up on treatment where additional serum and clinical data will be collected. The first visit will be 3 months after receiving the diagnosis and the second visit 6-12 months after the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects age 15-25 years
* Signed written informed consent

Exclusion Criteria:

* Less than 1 years from onset of menarche
* Use of hormonal contraceptives
* Documented ongoing pregnancy
* Major ovarian abnormalities, including subject with only one ovary, cysts and solid masses > 2 cm as detected by transvaginal ultrasound
* Malignancy ( documented malignancy, documentation of current radiation therapy or chemotherapy in medical record)

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Subjects who were assigned female at birth and are currently registered as females.
Study Population: Adolescent and young adult women aged between the ages of 15 and 25 with and without PCOS who present at the Women's Clinic of the University Hospital Erlangen.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The validation of new potential biomarkers for aid in the diagnoisis of PCOS in adolescent and young adult women | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Dittrich, Prof., Principal Investigator — University Hospital Erlangen
Locations (1):
- Department of Obstetrics and Gynecology, University Erlangen Hospital, Friedrich Alexander University of Erlangen-Nuremberg, Erlangen, Germany, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided